CLINICAL TRIAL: NCT04531176
Title: An ObEsity-centric Approach With and Without Anti-obesity Medications ComPared to the Usual-care ApprOach to Management of Patients With Obesity and Type 2 Diabetes in an Employer Setting: A Pragmatic Randomized Controlled Trial
Brief Title: EMI-EHP Weight Management and Type 2 Diabetes Pragmatic Trial
Acronym: EMPOWER-T2D
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: After an unplanned yet IRB approved interim analysis, it was found that there was not a significant difference between the 3 arms of the study. The study was closed due to futility. All Patients are off study and this study will not resume.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Bartolome Burguera, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-648
Record Dates: First submitted 2020-08-10; First posted 2020-08-28 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Phentermine; Naltrexone; Liraglutide; Orlistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Obesity-centric approach + AOM (Experimental): Participants will receive Cleveland Clinic's Integrated Medical WMP with medication for chronic weight management (Rx) for approximately two years. After discussing with the study doctor, participants will receive one of the following listed 4 drugs approved by the Food and Drug Administration (FDA) for long-term weight loss: 1) orlistat, 2) phentermine/topiramate extended-release, 3) naltrexone/bupropion extended-release and 4) liraglutide 3.0 mg
  Interventions: Other: Weight Management Program (WMP); Drug: Phentermine / Topiramate Extended Release Oral Capsule; Drug: naltrexone/bupropion extended-release; Drug: liraglutide 3.0 mg; Drug: Orlistat
- Obesity-centric approach without AOM (Experimental): Participants will receive Cleveland Clinic's Integrated Medical WMP alone for approximately two years.
  Interventions: Other: Weight Management Program (WMP)
- Usual care approach (Comorbidity-centric approach) (Active Comparator): Participants will receive the traditional usual care/standard of care approach to T2D, hypertension, hypercholesterolemia management for approximately two years.
  Interventions: Other: Traditional care

INTERVENTIONS:
Other: Weight Management Program (WMP) — Weight Management Program (WMP)
  Arms: Obesity-centric approach + AOM; Obesity-centric approach without AOM
Other: Traditional care — Traditional care
  Arms: Usual care approach (Comorbidity-centric approach)
Drug: Phentermine / Topiramate Extended Release Oral Capsule — Medication for chronic weight management (Rx)
  Arms: Obesity-centric approach + AOM
Drug: naltrexone/bupropion extended-release — Medication for chronic weight management (Rx)
  Arms: Obesity-centric approach + AOM
Drug: liraglutide 3.0 mg — Medication for chronic weight management (Rx)
  Arms: Obesity-centric approach + AOM
Drug: Orlistat — Medication for chronic weight management (Rx)
  Arms: Obesity-centric approach + AOM

SUMMARY:
This is a pragmatic, 24 month, single-center, randomized, open-label, parallel-group trial comparing an obesity-centric approach with a medically-supervised and comprehensive weight loss program (Cleveland Clinic's Endocrinology and Metabolism Institute's Integrated Weight Management Program) augmented by AOMs, vs. an obesity-centric approach with a medically-supervised and comprehensive weight loss program without AOMs, vs. the current usual care approach to general health management.

Informed consent will be obtained. IRB approval of the study will be obtained. 300 subjects (employees or spouses covered by our EHP) will be randomized 1:1:1 to receive either an obesity-centric approach with AOM therapy (N=100), an obesity-centric approach without AOM therapy (N=100), or the current usual care approach to general health management (N=100).

DETAILED DESCRIPTION:
Obesity affects nearly 40% of adults in the US and it is responsible for important medical problems including hypertension, dyslipidemia, T2D, depression, coronary heart disease, stroke, osteoarthritis, obstructive sleep apnea (OSA), fatty liver disease, and some cancers, to name a few4,5.

Obesity is responsible for the development of T2D and hypertension in more than 90% and 50% of cases, respectively6-7. Also more than 70% of patients with obesity have dyslipidemia. The prevalence of depression in patients with obesity is more than 50% and obesity is responsible for causing osteoarthritis in more than 25% of the patients8. Also, in the adult population, the prevalence of OSA is estimated to be ~25%, and as high as 45% in subjects with obesity9.

Patients with obesity have an increased risk of all-cause and cardiovascular death. In recognition of the biologic basis and seriousness of obesity, several professional health associations and organizations worldwide recognize obesity as a disease10.

Even though there is clear evidence in the literature that weight loss is associated with a dramatic improvement of obesity-related comorbidities and the patient's quality of life, in general, clinicians all over the world focus their attention on treating the diabetes, hypertension, hyperlipidemia and other comorbidities rather than the obesity itself, concentrating their efforts on improving blood glucose indices, blood pressure and LDL as well as triglycerides, and in many instances, prescribing anti-diabetes and antihypertensive medications that potentiate further weight gain11,12. As a result, clinicians are faced with a rising epidemic of obesity, perpetuating a preexisting epidemic of diabetes, hypertension, dyslipidemia, and metabolic syndrome.

Obesity is one of the biggest drivers of preventable chronic diseases and healthcare costs in the United States. Currently, estimates for these costs are $210 billion per year. In addition, obesity is associated with job absenteeism and with lower productivity while at work costing approximately $4.3 billion annually12,13.

As a person's BMI increases, so do the number of sick days, medical claims and healthcare costs. Individuals who suffer obesity spend 42% more on direct healthcare costs than adults who have a healthy weight. Individuals with grade 1 obesity (BMI between 30 and 35) are more than twice as likely as individuals with BMI < 30 to be prescribed prescription pharmaceuticals to manage medical conditions14.

Reducing obesity, improving nutrition, increasing physical activity, and making lifelong meaningful lifestyle changes can help lower costs through fewer doctor's office visits, tests, prescription drugs, sick days, emergency room visits and admissions to the hospital and lower the risk for a wide range of diseases.

A 2008 study by the Urban Institute, The New York Academy of Medicine and Trust for America's Health found that an investment of $10 per person in proven community-based programs to increase physical activity, improve nutrition, and prevent smoking and other tobacco use could save the country more than $16 billion annually within five years. That's a return of $5.60 for every $1 invested15.

In spite of these important facts there is a significant, yet much-underutilized role, for structured weight management programs, both with and without use of anti-obesity medications, to improve metabolic control for patients with obesity who have developed comorbidities such as hypertension hyperlipidemia and T2D. Unfortunately, these patients have a much higher risk of developing coronary artery disease and cancer.

The medical literature contains ample evidence which demonstrates the positive impact that a lifestyle intervention program augmented by FDA approved AOMs can have on anthropometric and metabolic parameters in patients with obesity who have developed significant comorbidities16-17. Lifestyle intervention, in the form of improving diet, eating behaviors and increasing physical activity, is first-line treatment for obesity and overweight, but the majority of people with obesity and overweight struggle to achieve and maintain their weight loss long-term. We hypothesize that an obesity-centric approach delivered through a medically-supervised and comprehensive weight loss program18, augmented by AOM, as the primary treatment of patients with obesity and T2D, will result in greater and sustainable weight loss, a better metabolic profile, (including glycemic blood pressure and cholesterol control) and improved quality of life (QOL) and treatment satisfaction when compared to an obesity-centric approach without AOM therapy or the current usual care/standard of care comorbidity-centric approach to general health management in patients with obesity and T2D. If confirmed, these findings would be expected to change our future approach to chronic diseases management, and reduce the rates of T2D, hypertension, and hyperlipidemia related complications (including heart disease and cancer) as well as the development of other obesity-related comorbidities, potentially reducing the long-term cost of care

ELIGIBILITY:
Inclusion Criteria:

1. Gender: men and women
2. Ethnicity: all ethnic groups
3. Age: ≥18, < 75 years
4. Diagnosis of T2D -A1C within the last 90 days must be >7.5%
5. Obesity, BMI ≥30
6. An Employee, or the significant other of an employee, that is covered by the Cleveland Clinic Employee Health Plan

Exclusion Criteria:

1. Type 1 diabetes or known latent autoimmune diabetes of adulthood (LADA)
2. Glomerular Filtration Rate <30 mL/min/1.73 m2 (calculated by the Chronic Kidney Disease Epidemiology Collaboration Equation, CKD-EPI)
3. Current glucocorticoid therapy
4. Currently or within the past 3 months receiving an anti-obesity medication, or any other medication used for the primary intent of weight loss
5. Any condition, unwillingness or inability, not covered by any of the other exclusion criteria, which, in the study clinician's opinion, might jeopardize the subject's safety or compliance with the protocol
6. Mental incapacity or language barrier
7. Pregnancy or plans to become pregnant within the next 2 years
8. Personal or family history of medullary thyroid carcinoma
9. Personal or family history of Multiple Endocrine Neoplasia syndrome type 2
10. History of acute pancreatitis, severe liver disease (Cirrhosis), or severe disease of digestive tract
11. History of congestive heart failure
12. History of bariatric or metabolic surgery/procedure
13. Visit with an endocrinologist within the past 1 year
14. Prior participation in the Endocrinology and Metabolism Institutes Integrated Weight Management Program

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2023-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bartolome Burguera, Principal Investigator — Institute Chairman
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Obesity-centric Approach + AOM | Obesity-centric Approach Without AOM | Usual Care Approach (Comorbidity-centric Approach)
Started | 24 | 26 | 24
Completed | 0 (Study was stopped early) | 0 (Study was stopped early) | 0 (Study was stopped early)
Not Completed | 24 | 26 | 24
Not completed — Study was stopped early | 24 | 26 | 24

BASELINE CHARACTERISTICS:
Population: Individual participants who were randomized to each arm of the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Obesity-centric Approach + AOM | Obesity-centric Approach Without AOM | Usual Care Approach (Comorbidity-centric Approach) | Total
Number analyzed (Participants) | 24 | 23 | 23 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 23 | 23 | 70
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53.5 [48.5 to 61.5] | 53.5 [47 to 60] | 53 [47.75 to 58.25] | 53.5 [47 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 13 | 41
  Male | 9 | 10 | 10 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 2 | 6
  Not Hispanic or Latino | 20 | 22 | 20 | 62
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 7 | 20
  White | 16 | 16 | 16 | 48
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 23 | 23 | 70

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Body Weight Between Baseline and 12 Months
Description: All relevant time points used in the calculation in the Time Frame between baseline and 12 months. Measured in the mean Change in body weight between baseline and 12 months measured in percentage (%) of body weight loss
Time Frame: 12 Months
Measure: Mean (90% Confidence Interval); unit: % of body weight
Arm/Group | Obesity-centric Approach + AOM | Obesity-centric Approach Without AOM | Usual Care Approach (Comorbidity-centric Approach)
Number analyzed (Participants) | 23 | 23 | 24
% of body weight | -8.74 [-10.74 to -6.74] | -6.68 [-8.71 to -4.65] | -4.48 [-6.52 to -2.45]
Statistical Analysis 1: Comparison: Obesity-centric Approach + AOM vs Obesity-centric Approach Without AOM vs Usual Care Approach (Comorbidity-centric Approach); Test type: Non-Inferiority — The results of non-inferiority test results are between pairwise groups. Non-inferiority was tested at the 0.05 level at 1 year and performed pairwise with Bonferroni adjusted significance levels for each paired comparison; p = 0.004, t-test, 1 sided — The non-inferiority regions were set to be 1% for weight loss change. When both primary endpoints are non-inferior, superiority testing at the 0.025 overall error level with Bonferroni adjustment for each endpoint at 1 year was then performed

2. Primary Outcome: Mean Change in A1C
Description: All relevant time points used in the calculation in the Time Frame between baseline and 12 months. Measured in the mean change of the percentage of glycosylated hemoglobin from baseline to 12 months
Time Frame: 12 Months
Measure: Mean (90% Confidence Interval); unit: Percentage of glycosylated hemoglobin
Arm/Group | Obesity-centric Approach + AOM | Obesity-centric Approach Without AOM | Usual Care Approach (Comorbidity-centric Approach)
Number analyzed (Participants) | 24 | 23 | 23
Percentage of glycosylated hemoglobin | -2.18 [-2.61 to -1.74] | -2.22 [-2.65 to -1.79] | -1.65 [-2.09 to -1.22]
Statistical Analysis 1: Comparison: Obesity-centric Approach + AOM vs Obesity-centric Approach Without AOM vs Usual Care Approach (Comorbidity-centric Approach); Test type: Non-Inferiority — Non-inferiority was tested at the 0.05 level at 1 year and performed pairwise with Bonferroni adjusted significance levels for each paired comparison; p = 0.05, t-test, 1 sided — The non-inferiority regions were set to be 0.5% for A1C. When both primary endpoints are non-inferior, superiority testing at the 0.025 overall error level with Bonferroni adjustment for each endpoint at 1 year was then performed

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Obesity-centric Approach + AOM | Obesity-centric Approach Without AOM | Usual Care Approach (Comorbidity-centric Approach)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/23 | 0/23
Other Adverse Events (participants affected / at risk) | 3/24 | 0/23 | 2/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obesity-centric Approach + AOM (N=24) | Obesity-centric Approach Without AOM (N=23) | Usual Care Approach (Comorbidity-centric Approach) (N=23)
Nausea, Vomiting, Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obesity-centric Approach + AOM (N=24) | Obesity-centric Approach Without AOM (N=23) | Usual Care Approach (Comorbidity-centric Approach) (N=23)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT04531176/Prot_SAP_001.pdf